CLINICAL TRIAL: NCT02675218
Title: Bone MicroArchitecture Abatacept in Rheumatoid Arthritis Patients (BMA2)
Brief Title: Bone MicroArchitecture Abatacept (BMA2)
Acronym: BMA2
Status: Terminated | Type: Observational
Why Stopped: No more inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1508203; 2015-005644-33 (EudraCT Number)
Record Dates: First submitted 2016-01-26; First posted 2016-02-05 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Doppler Effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be performed to determine the predictive value of joint inflammation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis.: Rheumatoid arthritis diagnosis according to ACR (American College of Radiology)/EULAR 2010 classification criteria.
  Interventions: Other: Patients with rheumatoid arthritis

INTERVENTIONS:
Other: Patients with rheumatoid arthritis — Doppler effect at 3 months after Abatacept treatment initiation.
  Other Names: Doppler effect

SUMMARY:
Rheumatoid Arthritis patients management reposes primarily on the use of disease-modifying antirheumatic drugs (DMARDs).

Among DMARDs available in 2015, researchers demonstrated the ability to reduce synovitis, biomarkers of inflammation, and bone destruction.

Given the demonstration of correlation between joint inflammation and structural progression at each joint level as well as the opportunity for bone remodeling with resolution of joint inflammation, researchers expect to observe an improvement in bone micro-architecture parameters specifically in rheumatoid arthritis patients without remaining joint inflammation 3 months following abatacept treatment initiation.

DETAILED DESCRIPTION:
Rheumatoid Arthritis patients management reposes primarily on the use of disease-modifying anti-rheumatic drugs. In patients responding insufficiently to Methotrexate, and/or other disease-modifying anti-rheumatic drugs (DMARD) strategies, with or without glucocorticoids, biological DMARD (TNF inhibitors, abatacept or tocilizumab, and, under certain circumstances, rituximab) should be commenced with Methotrexate. Among DMARD available in 2015, abatacept has demonstrated the ability to reduce synovitis, biomarkers of inflammation, and bone destruction. Monitoring rheumatoid arthritis patients after starting abatacept by US exams observed a strong reduction of power Doppler ultra-sonography at 3 months in two third of patients.

Given the demonstration of correlation between joint inflammation and structural progression at each joint level as well as the opportunity for bone remodeling with resolution of joint inflammation, researchers expect to observe an improvement in bone micro-architecture parameters specifically in rheumatoid arthritis patients without remaining joint inflammation 3 months following abatacept initiation.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form,
* Age ≥ 18 years,
* Rheumatoid arthritis diagnosis according to ACR/EULAR 2010 criteria
* Abatacept therapy sub-cutaneous required according EULAR recommendations
* Patients affiliated to health insurance

Exclusion Criteria:

* Other arthritis than rheumatoid arthritis,
* Contraindication to abatacept,
* Concomitant treatment with zoledronic acid (Aclasta®) or denosumab (Prolia®),
* Injection intravenously or intra-articular at the 2nd and 3rd metacarpophalangeal joint of the dominant hand during the 3 months prior to inclusion,
* Prior or planned joint surgery at the 2nd or 3rd metacarpophalangeal joint of the dominant hand over the one year study,
* No recent used of high density contrast material,
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients diagnosed according to ACR/EULAR 2010 criteria, and Abatacept therapy sub-cutaneous required according EULAR recommendation.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Value of joint inflammation | 1 year
  The predictive value of persistent joint inflammation on volumetric trabecular bone density is measured by high resolution pQCT (peripheral Quantitative Computed Tomography) after 1 year treatment with Abatacept.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (5):
- France (5):
  - Hôpital Édouard Herriot, Lyon
  - Ch Regional D'Orleans, Orléans
  - Assistance Publique-Hopitaux de Paris, Paris
  - Chu Saint Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No